CLINICAL TRIAL: NCT06913270
Title: Efficacy of Virtual Reality as an Adjunct for Procedural Pain and Anxiety Management in Burn Wound Care: A Single-Center, Randomized Controlled Trial
Brief Title: Virtual Reality Adjunct for Procedural Pain and Anxiety Management in Burn Wound Care
Acronym: VR-Burn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRBURN2025-01
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Burns; Burn Wound; Procedural Pain; Anxiety Acute
MeSH Terms: conditions — Burns; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel arms evaluating two distraction strategies during burn dressing changes.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the participants' group assignments. Participants, care providers, and investigators will be aware of the intervention received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Distraction (Experimental): Participants in this arm will receive standard analgesic care according to institutional protocols plus an immersive virtual reality (VR) distraction intervention. During each burn dressing change, participants will wear a head-mounted display delivering an interactive, engaging virtual environment specifically designed for distraction. This arm aims to assess the efficacy of VR in reducing procedural pain intensity and anxiety compared to the control condition.
  Interventions: Behavioral: Immersive Virtual Reality Distraction (IVRD)
- Nature Video Distraction (Active Comparator): Participants in this arm will receive the same standard analgesic care as the experimental group and will be provided with a non-VR distraction intervention. They will watch a nature video displayed on a tablet device during each burn dressing change session. This comparator is designed to control for the effects of distraction, allowing assessment of whether immersive VR provides additional benefit beyond conventional video distraction.
  Interventions: Behavioral: Nature Video Distraction (NVD)

INTERVENTIONS:
Behavioral: Immersive Virtual Reality Distraction (IVRD) — Intervention Description:
  Participants assigned to this intervention will receive standard analgesic care per institutional protocol in addition to an immersive virtual reality (VR) distraction intervention. During each burn dressing change, participants will wear a head-mounted display (HMD) that delivers an interactive and engaging virtual environment designed specifically to distract from procedural pain and reduce anxiety. The VR session will last for the entire duration of the dressing change (approximately 10-15 minutes) and will be administered during every session. The VR system is calibrated to provide high levels of sensory immersion to effectively divert attention from painful stimuli.
  Arms: VR Distraction
Behavioral: Nature Video Distraction (NVD) — Intervention Description:
  Participants in this intervention will receive the same standard analgesic care provided to all subjects and, in addition, will watch a nature video on a tablet device during the burn dressing change. The video distraction serves as an active comparator to the immersive VR. The nature video is selected to be calming and engaging, and it will be played continuously during the dressing change session (approximately 10-15 minutes). This intervention allows evaluation of whether immersive VR provides additional benefit in reducing procedural pain and anxiety over a standard video distraction.
  Arms: Nature Video Distraction

SUMMARY:
This randomized controlled trial is designed to evaluate the efficacy of immersive virtual reality (VR) as an adjunct to standard analgesia during dressing changes in adult burn patients. The study compares an intervention group receiving standard care combined with an immersive VR distraction (using a head-mounted display displaying an engaging virtual environment) versus a control group receiving standard care plus non-VR distraction (watching a nature video on a tablet). The primary outcomes include procedural pain intensity measured by the Visual Analog Scale (VAS) and anxiety levels measured by the State-Trait Anxiety Inventory (STAI). Secondary outcomes include patient satisfaction and physiological parameters (heart rate and blood pressure) recorded during the procedure. This trial addresses the critical gap of heterogeneity and small sample sizes noted in previous VR studies for burn care pain management (Dascal et al., 2017).

DETAILED DESCRIPTION:
Procedural pain during dressing changes for burn wound care remains a substantial clinical challenge affecting both patient comfort and treatment compliance. Immersive VR technology has been suggested as an effective distraction technique, potentially reducing pain and associated anxiety by providing a highly engaging alternative sensory input. However, previous studies have been limited by variable protocols and modest sample sizes.

In this single-center RCT, adult burn patients aged 18-65 years with partial-thickness burns scheduled for routine dressing changes will be enrolled. Participants will be randomly assigned in a 1:1 ratio to either:

Intervention Group: Standard care (analgesia as per institutional protocol) plus immersive VR distraction (using a commercially available head-mounted display with interactive virtual environments) Control Group: Standard care plus non-VR distraction, operationalized as watching a nature video on a tablet device.

Randomization will be computer generated.

Outcome assessors will be blinded to treatment assignment. The primary outcome measures are procedural pain intensity (assessed using a 10-cm Visual Analog Scale immediately post-procedure) and anxiety (assessed using the State-Trait Anxiety Inventory immediately post-procedure). Secondary endpoints include patient-reported satisfaction with the distraction modality and objective physiological parameters (heart rate and blood pressure) monitored throughout the procedure.

Data will be collected at each dressing change session over the study period, and repeated measures analysis will be applied to assess between-group differences.

ELIGIBILITY:
Inclusion Criteria:

Adult burn patients (18-65 years) with confirmed partial-thickness burns. Scheduled for routine dressing changes. Able to provide informed consent. Baseline pain score of ≥4/10 during a dressing change session.

Exclusion Criteria:

Patients with cognitive impairment preventing comprehension of the intervention.

History of severe motion sickness or visual impairments that preclude the use of VR devices.

Patients with contraindications to standard analgesic care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-12 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Functional Status via Burn Specific Health Scale - Brief (BSHS-B) | Assessments will be conducted at baseline (within 2 weeks post-discharge) and at follow-up visits at 3, 6, and 12 months.
  The Burn Specific Health Scale - Brief (BSHS-B) is a validated questionnaire designed to assess physical, psychosocial, and functional outcomes in burn survivors. It evaluates domains such as physical functioning, pain, emotional health, and social reintegration. Changes in functional status over time will help determine the impact of the burn injury and the effect of the intervention on recovery.
Return-to-Work Rate | Assessed at 12 months post-discharge.
  This outcome measure evaluates the proportion of participants who have successfully returned to work at 12 months post-discharge. Return-to-work status will be verified by self-report and cross-referenced with available medical and employment records, serving as an indicator of long-term functional recovery and social reintegration.

SECONDARY OUTCOMES:
Quality of Life (QoL) via SF-36 Health Survey | Evaluations will occur at baseline (within 2 weeks post-discharge) and at 3, 6, and 12 months follow-up.
  The SF-36 Health Survey is a comprehensive, validated instrument designed to measure quality of life across eight domains, including physical functioning, bodily pain, general health perceptions, vitality, social functioning, role limitations due to physical and emotional problems, and mental health. This will provide insight into the broader impact of burn injuries and recovery over time.
Range of Motion (ROM) Measurements | Measurements will be recorded at baseline and at follow-up visits at 3, 6, and 12 months.
  Range of motion (ROM) in the affected areas will be assessed using standardized goniometry. This measurement quantifies physical mobility and joint function, providing objective data on the physical recovery and potential functional limitations post-burn injury.
Psychological Well-Being via Hospital Anxiety and Depression Scale (HADS) | HADS assessments will be administered at baseline (within 2 weeks post-discharge) and then at 3, 6, and 12 months follow-up.
  The Hospital Anxiety and Depression Scale (HADS) is a validated self-report questionnaire used to assess anxiety and depressive symptoms. Improving psychological well-being is a key aspect of overall recovery for burn survivors.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No